CLINICAL TRIAL: NCT05361759
Title: National Tunisian Registry of Cardiac Implantable Electronic Devices (NATURE-CIED)
Brief Title: National Tunisian Registry of Cardiac Implantable Electronic Devices
Acronym: NATURE-CIED
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society of Cardiology and Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: DAC-012-NATURECIED
Record Dates: First submitted 2022-04-30; First posted 2022-05-05 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Implantable Electronic Devices
Keywords: Cardiac Implantable Electronic Devices; Heart; Pacemaker; Implantable Cardioverter Defibrillator; Cardiac Loop Recorders; Biventricular Pacemakers; Heart rhythm disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cardiac Implantable Electronic Devices — Description of Cardiac Implantable Electronic Devices

SUMMARY:
The National Tunisian Registry of Cardiac Implantable Electronic Devices is an observational, prospective and multicenter study aiming to assess the epidemiological, clinical and therapeutic profile of cardiac implantable electronic Devices in Tunisia. Cardiologists from both sectors (public and private) are participating in the study, with 26 investigational centers. Data is captured electronically by DACIMA Clinical Suite, according to FDA 21 CFR part 11 (Food and Drug Administration 21 Code of Federal Regulations part 11), HIPAA (Health Insurance Portability and Accountability Act) & ICH (International Conference on Harmonisation) requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients originated from Tunisia
* Signed informed consent
* Patients undergoing a cardiac implantable electronic device procedure

Exclusion Criteria:

* Informed Consent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac implantable electronic device procedure
Sampling Method: Non-Probability Sample
Enrollment: 1518 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of patients undergoing cardiac implantable electronic devices in Tunisia | at inclusion
  Number of subjects with heart disease (heart failure, rythm disorder) and willing to participate at the study and who are eligible for cardiac implantable electronic devices procedures

SECONDARY OUTCOMES:
Heart complication | at 12 months of follow-up
  Number of patients with cardiovascular event, including death, tamponade, pericarditis, heart failure, worsening of valvular disease, moving the right ventricular lead, compartment infection, phrenic stimulation, conductor breakage, or any other cardiovascular complication related to the cardiac implantable electronic device

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Chabrak, MD, Study Chair — Tunisian Society of Cardiology and Cardiovascular Surgery; Abdeddayem Haggui, MD, Study Director — Tunisian Society of Cardiology and Cardiovascular Surgery; Salma Krichène, MD, Principal Investigator — Tunisian Society of Cardiology and Cardiovascular Surgery; Slim Kacem, MD, Principal Investigator — Tunisian Society of Cardiology and Cardiovascular Surgery; Sonia Marrakchi, MD, Principal Investigator — Tunisian Society of Cardiology and Cardiovascular Surgery; Emna Allouche, MD, Principal Investigator — Tunisian Society of Cardiology and Cardiovascular Surgery
Locations (1):
- The Tunisian Society of Cardiology and CardioVascular Surgery, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chabrak S, Haggui A, Allouche E, Ouali S, Ben Halima A, Kacem S, Krichen S, Marrakchi S, Fehri W, Mourali MS, Jabbari Z, Ben Halima M, Neffati E, Heraiech A, Slim M, Kachboura S, Gamra H, Hassine M, Kraiem S, Kammoun S, Bezdah L, Jridi G, Bouraoui H, Kammoun S, Hammami R, Chettaoui R, Ben Ameur Y, Azaiez F, Tlili R, Battikh K, Ben Slima H, Chrigui R, Fazaa S, Sanaa I, Ellouz Y, Mosrati M, Milouchi S, Jarmouni S, Ayadi W, Akrout M, Razgallah R, Neffati W, Drissa M, Charfeddine S, Abdessalem S, Abid L, Zakhama L. National Tunisian Study of Cardiac Implantable Electronic Devices: Design and Protocol for a Nationwide Multicenter Prospective Observational Study. JMIR Res Protoc. 2024 Apr 8;13:e47525. doi: 10.2196/47525. PMID 38588529
- See also: Tunisian Society of Cardiology and Cardiovascular Surgery Website — http://www.stcccv-tunisie.com/